CLINICAL TRIAL: NCT07146724
Title: The Effects of Pilates-Based Exercises on Hamstring Flexibility, Plantar Pressure Sensation, and Dynamic Balance
Brief Title: The Effects of Pilates-based Exercises on the Posterior Leg Muscles
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, asuman saltan, Principal Investigator, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/187
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-03

CONDITIONS: Exercise Therapy
Keywords: Pilates, Exercise Therapy, Randomized Controlled Trial
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ınterventıon arm (Active Comparator): Pilates-Based Exercise Group
  Interventions: Other: Exercise
- control arm (No Intervention): Control Group (No Exercise Intervention)

INTERVENTIONS:
Other: Exercise — The intervention consists of a pilates-based exercise program specifically designed to target hamstring flexibility, plantar pressure sensitivity, and dynamic balance.
  Unlike general fitness-oriented pilates, this program includes a combination of mat-based and functional pilates movements adapted to improve posterior chain flexibility and sensory feedback in the lower extremities.
  The protocol includes 3 sessions per week for 8 weeks - 1 session conducted face-to-face under physiotherapist supervision and 2 sessions as a monitored home exercise. Exercise progression is standardized, and all sessions follow a validated physiotherapy protocol tailored for university-aged individuals with clinically measured hamstring shortening.
  Arms: ınterventıon arm

SUMMARY:
This randomized controlled study aims to investigate the effects of a pilates-based exercise program on hamstring flexibility, plantar pressure sensation, and dynamic balance in university students aged 18 to 24 years.

Participants diagnosed with hamstring tightness through the Sit and Reach test will be randomly assigned to an exercise group and a control group. The intervention group will undergo an 8-week pilates-based home and supervised exercise program. Outcomes will be evaluated before and after the intervention using Sit and Reach, monofilament sensory testing, and the Y Balance Test.

The study seeks to identify whether a non-invasive physical activity like pilates can improve neuromuscular and sensory parameters in young adults.

ELIGIBILITY:
Inclusion Criteria:Aged between 18-24 years

Enrolled students at Yalova University

Diagnosed with hamstring shortening (measured via Sit and Reach Test)

Willing to participate voluntarily and provide informed consent

Not currently participating in any regular exercise program -

Exclusion Criteria:Diagnosed with hypermobility syndrome

History of orthopedic surgery in the lower extremities in the past 6 months

Neurological or musculoskeletal diseases affecting mobility

Having systemic chronic disease (e.g., diabetes, MS)

Currently under physiotherapy or similar treatment

Unwilling or unable to follow the 8-week intervention schedule

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Hamstring Flexibility | 8 weeks
  Hamstring flexibility will be measured using the Sit and Reach Test. Participants will perform the test at baseline and at the end of the 8-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova University faculty of health science department of physiotherapy and rehabilitation, Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No